CLINICAL TRIAL: NCT04973813
Title: Effects of an Active Choice Intervention on Physical Activity Intentions and Behaviour Among Physically Inactive Adults: A Four-Arm Web-Based Experiment
Brief Title: Active Choice Intervention About Physical Activity for Physically Inactive Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Amsterdam UMC, location VUmc (Other)
Responsible Party: Principal Investigator, Lorraine Landais, Principal Investigator, Amsterdam UMC, location VUmc
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 2020.142
Record Dates: First submitted 2021-06-11; First posted 2021-07-22 (Actual); Last update posted 2021-07-22 (Actual); Status verified 2021-07

CONDITIONS: Physical Activity
Keywords: Physical activity intervention; Active choice; Decision making; Web-based
MeSH Terms: conditions — Motor Activity | interventions — Guidelines as Topic

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Guideline + Active Choice + action&coping planning (GA+) (Experimental): Participants received a web-based intervention consisting of information (including the national physical activity guideline) and several assignments. Assignments included: completing a decision balance sheet; indicating the importance of personal values and the time, effort and energy spent on these personal values; action planning; identifying barriers to physical activity; coping planning.
  Interventions: Behavioral: Guideline + Active Choice + action&coping planning (GA+)
- Guideline + Active Choice (GA) (Experimental): Participants received a web-based intervention consisting of information (including the national physical activity guideline) and several assignments. Assignments included: completing a decision balance sheet; indicating the importance of personal values and the time, effort and energy spent on these personal values; identifying barriers to physical activity.
  Interventions: Behavioral: Guideline + Active Choice (GA)
- Guideline + Information (GI) (Experimental): Participants received the national physical activity guideline, and information about pros and cons of physical activity, and possible barriers to physical activity.
  Interventions: Behavioral: Guideline + information (GI)
- Guideline (G) (Other): Comparison arm. Participants received the national physical activity guideline.
  Interventions: Behavioral: Guideline (G)

INTERVENTIONS:
Behavioral: Guideline + Active Choice + action&coping planning (GA+) — Web-based intervention consisting of information and assignments, including: completing a decision balance sheet; indicating the importance of personal values and the time, effort and energy spent on these personal values; action planning; identifying barriers to physical activity; coping planning
  Arms: Guideline + Active Choice + action&coping planning (GA+)
Behavioral: Guideline + Active Choice (GA) — Web-based intervention consisting of information and several assignments, including: completing a decision balance sheet; indicating the importance of personal values and the time, effort and energy spent on these personal values; identifying barriers to physical activity.
  Arms: Guideline + Active Choice (GA)
Behavioral: Guideline + information (GI) — Web-based information about the national physical activity guideline, pros and cons of physical activity, and possible barriers to physical activity.
  Arms: Guideline + Information (GI)
Behavioral: Guideline (G) — Web-based information about the national physical activity guideline.
  Other Names: Comparison arm
  Arms: Guideline (G)

SUMMARY:
This web-based experimental study aims to ascertain whether promoting an active (i.e. conscious and autonomous) choice process about physical activity results in better behavioural outcomes (e.g. physical activity) and psychological outcomes (e.g. physical activity intention) compared to promoting a passive choice process in physically inactive adults.

DETAILED DESCRIPTION:
In this web-based experimental study, the investigators will use a pre-test post-test four-arm parallel design to compare the effect of promoting an active choice process versus a passive choice process about physical activity on behavioural outcomes (e.g. physical activity behaviour, perceived increase in physical activity) and psychological outcomes (e.g. physical activity intention, commitment) among physically inactive adults.

Participants will be randomized to one of four groups. Participants in group GA+ will be encouraged to make a very active choice by weighing advantages and disadvantages of physical activity, considering personal values, identifying barriers and engaging in action and coping planning. The intervention for group GA is similar, but lacks the action and coping planning exercises. In the other two groups, a passive choice process will be promoted by only providing information: Group G will read the national physical activity guideline and group GI will read the guideline and information about possible advantages and disadvantages and barriers to physical activity. Behavioural and psychological outcomes will be assessed at the first measurement and follow-up measurement. Regression analyses will be performed to examine intergroup differences. In addition, sensitivity analyses and a process evaluation will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Low levels of physical activity (i.e. physically active for at least 30 minutes on <5 days a week and engaging in <150 minutes of physical activity in total throughout an average week)

Exclusion Criteria:

* Pregnancy
* Wheelchair user
* Not being able to walk a minimum of 100 meters

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 564 (Actual)
Dates: Start 2020-09-04 (Actual); Primary Completion 2020-10-09 (Actual); Study Completion 2020-10-09 (Actual)

PRIMARY OUTCOMES:
Intention | Directly after the intervention (Day 0)
  Intention to become more physically active (yes/no), assessed by a questionnaire
Physical activity | Change from baseline at approximately 18 days
  Physical activity levels (MET minutes per week), assessed by the short form of the International Physical Activity Questionnaire (IPAQ)

SECONDARY OUTCOMES:
Sitting time | Change from baseline at approximately 18 days
  Sitting time (minutes per day), assessed by the short form of the International Physical Activity Questionnaire (IPAQ)
Perceived change in physical activity compared to baseline | Change from baseline at approximately 18 days
  Questionnaire item: Participants' self-perceived change in physical between baseline and follow-up. Dichotomous outcome (change/no change).
Intention strength | Change from day 0, at approximately 18 days
  Questionnaire item: scale 0 (no strong intention) - 10 (very strong intention). a higher score indicates higher intention strength.
Active choice | Directly after the intervention (Day 0)
  Degree to which an active choice is made; a composite score of 9 items on a scale of 1 (totally not agree) - 5 (totally agree); a higher score indicates a more active choice.
Autonomous choice | Directly after the intervention (Day 0)
  Degree to which an autonomous choice is made; 2 items on a scale of 1 - 10. For the first item, a higher score indicates a more autonomous choice, whereas for the second item, a higher score indicates a less autonomous choice.
Commitment | Directly after the intervention (Day 0)
  Commitment to become more physically active; 1 item on a scale of 0 (no commitment) - 10 (high commitment). A higher score indicates higher commitment.
Commitment | Change from day 0, at approximately 18 days follow-up
  Commitment to become more physically active; 1 item on a scale of 0 (no commitment) - 10 (high commitment). A higher score indicates higher commitment.
Self-efficacy | Directly after the intervention (Day 0)
  Self-efficacy to become more physically active; 2 items on a scale of 1 (no self-efficacy) - 10 (high self-efficacy). A higher score indicates more self-efficacy.
Self-efficacy | Change from day 0, at approximately 18 days follow-up
  Self-efficacy to become more physically active; 2 items on a scale of 1 (no self-efficacy) - 10 (high self-efficacy). A higher score indicates more self-efficacy.
Satisfaction about one's plan | Directly after the intervention (Day 0)
  Degree of satisfaction with one's plan to become or not become more physically active on a scale of 1 (no satisfaction) to 10 (high satisfaction).
Alignment of choice with personal values | Directly after the intervention (Day 0)
  Extent to which one's plan to become/ not become more physically active corresponds with what one considers important; 1 item on a scale of 1 (no alignment) - 10 (high alignment)
Perceived advantages and disadvantages of physical activity | During intervention (Day 0)
  Open-ended questions about the perceived advantages and disadvantages of one's current physical activity behavior, and of increasing physical activity.
Value of health | During intervention (Day 0)
  Importance of the value 'health', on a scale of 1 (not important at all) to 10 (very important), and the time, effort and energy spent on health on a scale of 1 (no time, effort and energy) to 10 (very much time, effort and energy)
Values influencing physical activity | During intervention (Day 0)
  The extent to which the following values impact one's physical activity levels on a scale of 1 (no influence) to 10 (high influence): responsibility, achievement, pleasure, family, friendships, balance.
Plans to change physical activity | During intervention (Day 0)
  Open-ended questions about the preferred kind of physical activity, frequency, location, days and start date.
Perceived barriers to physical activity | During intervention (Day 0)
  Open-ended question asking about perceived barriers to physical activity
Plans to cope with perceived barriers | During intervention (Day 0)
  Open-ended questions about the ways one could cope with each perceived barriers
Factors supporting physical activity | Follow-up; approximately 18 days after the intervention (day 0)
  Question about the factors that supported or would support physical activity. Multiple choice question.
Barriers to physical activity | Follow-up; approximately 18 days after the intervention (day 0)
  Question about the barriers that hindered physical activity in the past two weeks. Multiple choice question.

CONTACTS AND LOCATIONS:
Overall Officials: Danielle Timmermans, Prof. dr., Study Director — Amsterdam UMC; Evert Verhagen, Prof. dr., Study Director — Amsterdam UMC
Locations (1):
- VUMedicalCenter, Amsterdam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
We plan to make all anonymized data available during publication, e.g. via clinicaltrials.gov.
Supporting Information: Study Protocol, SAP
Time Frame: Data will become available during publication.
Access Criteria: No access restrictions.

REFERENCES:
- [Derived] Landais LL, Jelsma JGM, Verhagen EALM, Timmermans DRM, Damman OC. Awareness of a disconnect between the value assigned to health and the effort devoted to health increases the intention to become more physically active. Health Psychol Behav Med. 2023 Jul 30;11(1):2242484. doi: 10.1080/21642850.2023.2242484. eCollection 2023. PMID 37529054
- [Derived] Landais LL, Damman OC, Jelsma JGM, Verhagen EALM, Timmermans DRM. Promoting an active choice among physically inactive adults: a randomised web-based four-arm experiment. Int J Behav Nutr Phys Act. 2022 Apr 27;19(1):49. doi: 10.1186/s12966-022-01288-y. PMID 35477419

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-06-29): https://cdn.clinicaltrials.gov/large-docs/13/NCT04973813/Prot_SAP_000.pdf